CLINICAL TRIAL: NCT01028378
Title: Topography-Guided LASIK Using the ALLEGRETTO WAVE Eye-Q 400 Hz Excimer Laser System For the Treatment of Manifest and Cornea Based Myopic and Hyperopic Optical Errors
Brief Title: Safety and Efficacy Study of Topography-Guided LASIK to Treat Myopia and Hyperopia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinical Research Consultants, Inc. (Industry)
Collaborators: Alcon Research (Industry); WaveLight AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-CAT-001
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topography-guided LASIK (Experimental): Topography-guided LASIK for Myopia or Hyperopia
  Interventions: Device: T-CAT topography-guided LASIK treatment with the Allegretto Wave Eye-Q 400 Hz Excimer Laser

INTERVENTIONS:
Device: T-CAT topography-guided LASIK treatment with the Allegretto Wave Eye-Q 400 Hz Excimer Laser

SUMMARY:
This purpose of this study is to evaluate the safety and effectiveness of a topography-based custom ablation treatment using the ALLEGRETTO WAVE® Eye-Q 400 Hz laser system for treating myopia and hyperopia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Signed Informed Consent;
* Willingness and ability to comply with schedule for follow-up visits;
* be a candidate for topography guided LASIK treatment of myopia or hyperopia in both eyes based on your doctors examination of your eyes;
* Intended treatment is targeted for emmetropia;
* Stable refraction (0.5 D or less change in manifest refraction spherical equivalent (MRSE) per year) for 12 months or longer, based on previous clinical records or prescription history (e.g., old glasses/contact lens prescriptions).
* Able to obtain a reliable corneal topography that can be used to determine the T-CAT treatment plan;
* Best spectacle-corrected visual acuity (BSCVA) 20/25 or better in each eye;
* Less than 0.75 D spherical equivalent (SE) difference between cycloplegic and manifest refractions.
* Is not a contact lens wearer or, if wearing contact lenses, has discontinued wearing contact lenses for the required period of time and completed the contact lens stability check;
* be able to maintain your eye position steady during the course of the treatment.

Exclusion Criteria:

* History of prior refractive treatment;
* Mixed astigmatism refractive error;
* Lenticular astigmatism that, in the investigator's opinion, is clinically significant;
* Corneal topography showing evidence of keratoconus, keratoconus suspect, forme fruste keratoconus, pellucid marginal degeneration, or other topographic abnormality that would place the eye at risk for developing post-refractive corneal ectasia;
* Treatment plan for T-CAT would predict a residual stromal bed thickness less than 250 microns;
* History or current evidence of corneal or other anterior segment disease that might reasonably be expected to affect the outcome of treatment (e.g., herpes simplex keratitis, herpes zoster keratitis, recurrent erosion syndrome, corneal melt, corneal dystrophy, etc.);
* Evidence of retinal vascular disease;
* Female patients who are pregnant or lactating or plan to become pregnant during the course of the study;
* A known sensitivity to study medications;
* Nystagmus or any other condition that would prevent a steady gaze during the LASIK treatment or other diagnostic tests;
* Corneal dystrophy or corneal guttae;
* Pathology involving the iris (e.g., coloboma, tears, cuts, significant pigment loss, etc.);
* Residual, recurrent or active ocular pathology;
* Previous intraocular or corneal surgery that might confound the outcome or increase the risk of the study;
* Acute or chronic illness that might increase the risk or confound the outcome of the study (e.g., diagnosed autoimmune disease, systemic connective tissue disease, clinically significant atopic disease, diabetes mellitus, etc.)
* The use of systemic medications that may confound the outcome or increase the risk of the study, including, but not limited to: corticosteroids and antimetabolites;
* Intraocular pressure > 23 mm Hg, a history of glaucoma, or a glaucoma suspect;
* An increased risk for developing strabismus after treatment (applicable only to treatment of hyperopic refractive errors);
* Presence or history of any other condition or finding that, in the investigator's opinion, makes the patient unsuitable as a candidate for LASIK or study participation or may confound the outcome of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doyle Stulting, M.D., Ph.D., Study Director — Woolfson Eye Institute/Medical Monitor
Locations (10):
- United States (10):
  - Milauskas Eye Institute, La Quinta, California
  - Gordon & Weiss Vision Institute, San Diego, California
  - Woolfson Eye Institute, Atlanta, Georgia
  - Emory Vision, Atlanta, Georgia
  - Bond Eye Associates, Peoria, Illinois
  - Durrie Vision, Overland Park, Kansas
  - TLC Laser Eye Center, Greensboro, North Carolina
  - Memorial Eye Institute, Harrisburg, Pennsylvania
  - Laser Vision of Texas, Houston, Texas
  - International Eye Care Laser Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Topography-guided LASIK: Topography-guided LASIK for Myopia or Hyperopia
  T-CAT topography-guided LASIK treatment with the Allegretto Wave Eye-Q 400 Hz Excimer Laser
Period: Overall Study
Arm/Group | Topography-guided LASIK
Started | 212 (212 participants (249 eyes) with myopia)
Completed | 195 (195 participants (230 eyes) with myopia)
Not Completed | 17
Not completed — Lost to Follow-up | 12
Not completed — Withdrawal by Subject | 1
Not completed — Adminstrative Reasons | 4

BASELINE CHARACTERISTICS:
Population: 212 participants (249 eyes)
Arm/Group | Topography-guided LASIK
Number analyzed (Participants) | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 119
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 157
  Black | 4
  Asian | 8
  Hispanic | 37
  Other | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Manifest Refraction Spherical Equivalent (MRSE) +/- 0.50 D
Time Frame: 12 month
Measure: Number (95% Confidence Interval); unit: Percentage of Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Topography-guided LASIK
Number analyzed (Participants) | 195
Number analyzed (Number of Eyes) | 230
Percentage of Eyes | 94.78 [91.8 to 97.7]

2. Primary Outcome: Percentage of Eyes With Manifest Refraction Spherical Equivalent (MRSE) +/- 1.00 D
Time Frame: 12 month
Measure: Number (95% Confidence Interval); unit: Percentage of Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Topography-guided LASIK
Number analyzed (Participants) | 195
Number analyzed (Number of Eyes) | 230
Percentage of Eyes | 99.57 [98.7 to 100]

3. Primary Outcome: Percentage of Eyes With Manifest Refraction Spherical Equivalent (MRSE) +/- 2.00 D
Time Frame: 12 month
Measure: Number (95% Confidence Interval); unit: Percentage of Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Topography-guided LASIK
Number analyzed (Participants) | 195
Number analyzed (Number of Eyes) | 230
Percentage of Eyes | 100 [100 to 100]

4. Primary Outcome: Percentage of Eyes With Uncorrected Visual Acuity (UCVA) 20/20 or Better
Time Frame: 12 month
Measure: Number (95% Confidence Interval); unit: Percentage of Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Topography-guided LASIK
Number analyzed (Participants) | 195
Number analyzed (Number of Eyes) | 230
Percentage of Eyes | 92.61 [89.2 to 96.1]

5. Primary Outcome: Percentage of Eyes With UCVA 20/40 or Better if BSCVA 20/20 or Better Preoperatively
Time Frame: 12 month
Measure: Number (95% Confidence Interval); unit: Percentage of Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Topography-guided LASIK
Number analyzed (Participants) | 195
Number analyzed (Number of Eyes) | 230
Percentage of Eyes | 99.56 [98.7 to 100]

6. Primary Outcome: Percentage of Eyes With Loss of 2 or More Lines Best Spectacle-Corrected Visual Acuity (BSCVA)
Time Frame: 12 month
Measure: Number (95% Confidence Interval); unit: Percentage of Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Topography-guided LASIK
Number analyzed (Participants) | 195
Number analyzed (Number of Eyes) | 230
Percentage of Eyes | 0.43 [0 to 1.3]

7. Primary Outcome: Percentage of Eyes With Best Spectacle-Corrected Visual Acuity (BSCVA) Worse Than 20/40
Time Frame: 12 month
Measure: Number (95% Confidence Interval); unit: Percentage of Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Topography-guided LASIK
Number analyzed (Participants) | 195
Number analyzed (Number of Eyes) | 230
Percentage of Eyes | 0 [0 to 0]

8. Primary Outcome: Percentage of Eyes With an Increase > 2D Cylinder (Spherical Only)
Time Frame: 12 month
Measure: Number (95% Confidence Interval); unit: Percentage of Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Topography-guided LASIK
Number analyzed (Participants) | 195
Number analyzed (Number of Eyes) | 230
Percentage of Eyes | 0 [0 to 0]

9. Primary Outcome: Percentage of Eyes With Best Spectacle-corrected Visual Acuity (BSCVA) Worse Than 20/40 if 20/20 or Better Preoperatively
Time Frame: 12 month
Measure: Number (95% Confidence Interval); unit: Percentage of Eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Topography-guided LASIK
Number analyzed (Participants) | 195
Number analyzed (Number of Eyes) | 230
Percentage of Eyes | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Topography-guided LASIK
Serious Adverse Events (participants affected / at risk) | 0/195
Other Adverse Events (participants affected / at risk) | 2/195
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topography-guided LASIK (N=195)
BSCVA loss of 2 or more lines (Eye disorders) | 1
Retinal Detachments (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No